CLINICAL TRIAL: NCT04489043
Title: Exercise, Prediabetes and Diabetes After Renal Transplantation.
Acronym: EXPRED
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Universitario de Canarias (Other)
Collaborators: Instituto de Salud Carlos III (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: EXPRED
Record Dates: First submitted 2020-07-15; First posted 2020-07-28 (Actual); Last update posted 2020-07-28 (Actual); Status verified 2020-07

CONDITIONS: Diabetes Mellitus
Keywords: PreDiabetes; Exercise; Late post transplant Diabetes Mellitus (PTDM); Renal transplantation
MeSH Terms: conditions — Diabetes Mellitus; Prediabetic State; Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Patients with prediabetes beyond 12 months after transplantation will be included. Prediabetes will be diagnosed based on fasting glucose levels and oral glucose tolerance tests (OGTT). Patients will be treated with a stepped training intervention, starting with an aerobic exercise training (brisk walking, swimming and cycling) 5 times per week, 30 min/day. Aerobic exercise training will gradually increase to 60 min/day or in combination with anaerobic exercise training in case of persistent prediabetes. The reversibility/persistence of prediabetes will be measured with fasting glucose and OGTTs at every 3 months.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exercise and healthy life style recommendations (Experimental): A planned exercise programme to test the impact of this treatment. An Oral Glucose Tolerant Test (OGTT) at intermediate time points in order to increase the frequency and duration of aerobic exercise and eventually to add anaerobic/resistance training.
  Interventions: Other: Exercise and healthy lifestyle recommendations

INTERVENTIONS:
Other: Exercise and healthy lifestyle recommendations — In the present study, renal transplant patients with proven prediabetes will do a planned exercise programme to test the impact of this treatment on the reversibility of prediabetes. Thus, the persistance of recurrency of prediabetes assessed by an Oral Glucose Tolerant Test (OGTT) at intermediate time points (3, 6 and 9 months) will be checked in order to increase the frequency and duration of aerobic exercise and eventually to add anaerobic/resistance training.

SUMMARY:
This study is designed to evaluate the feasibility of exercise to reverse prediabetes after transplantation to prevent Posttransplantation Diabetes Mellitus (PTDM).

DETAILED DESCRIPTION:
The hypothesis of the study is that exercise will promote the reversibility to normal glucose metabolism in patients with prediabetes and eventually reduce the incidence of PTDM in renal transplant. The main objective of the study is to induce the reversibility of prediabetes by means of exercise. Additionally, the secondary objectives are: (a) to evaluate the compliance of exercise (b) improvements in metabolic risk factors profile: obesity, triglycerides, blood pressure and HDL cholesterol.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years old.
* Renal transplantation: beyond 6-12 months after transplantation with stable renal function
* IFG: 100-125 mg/dl and IGT 140-199 mg/dl.
* Ability or capacity to perform exercise.

Exclusion Criteria:

* Clinical conditions that preclude the treatment with exercise i.e. clinical instability: active infection, cancer, acute cardiovascular disease, advanced renal disease, pulmonar hypertension, chronic obstructive pulmonary disease, severe reumatological disorders, arthrosis, arthritis limb amputation, etc.
* Inability to understand the protocol.
* Severe psychological disease.
* PTDM.
* Diabetes before transplantation.

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2019-09-05 (Actual); Primary Completion 2019-12-05 (Actual); Study Completion 2021-10-01 (Estimated)

PRIMARY OUTCOMES:
Oral glucose tolerance test (OGTT) | Baseline and 3 months-12 months, every 3 months
  After a 10-12 h overnight fast, a standard 75-g OGTT with samples taken at 0 min (glucose-insulin) and 120 minutes (glucose) will be performed at screening-baseline and after 3,6,9,12 months. Patients must be clinically stable without conditions that could induce transient hyperglycaemia or insulin resistance, i.e. infections, acute rejection, renal failure or cardiovascular disease. The presence of any of these conditions postponed the test for at least 3 months after full recovery. Also, serum and urinary samples will be taken and storage at -80 degrees.

SECONDARY OUTCOMES:
Compliance | Baseline and 3 months-12 months, every 3 months
  To ensure compliance, the following measures will be implemented: (a) contact by phone one time per week (at the end of the week) in the first 3 months up to the end of the study, (b) individual interview every month to reinforce lifestyle changes and follow all recommended in the exercise prescription; (c) the use of a gadget (xiaomi mi band) to see daily routines of patients and every training prescription; this analyses the time, frequency, burned calories, velocity and distance, among others, to reach the established goal by the physiotherapist.
Analitics | Baseline and 3 months-12 months, every 3 months
  To evaluate the improvements in metabolic risk factors profile: obesity, triglycerides, blood pressure and HDL cholesterol.hemogram (hematocrit, haemoglobin, white blood count), biochemist tests: creatinine, HbA1c, total, LDL and HDL cholesterol, triglycerides, uric acid, hepatic enzymes (ASAT, ALAT), levels of immunosuppression, albumin, creatinine, albuminuria, proteinuria in an isolated urinary samples.
Test the reversibility of prediabetes | Baseline and 3 months-12 months, every 3 months
  There is a n exercise programme to test the impact of this treatment on the reversibility of prediabetes. Thus, the persistance of recurrency of prediabetes assessed by an OGTT at intermediate time points (3, 6 and 9 months) will be checked in order to increase the frequency and duration of aerobic exercise and eventually to add anaerobic/resistance training.
Cardiorrespiratory fitness test | Baseline and 3 months-12 months, every 3 months
  Cardiopulmonary exercise testing (CPTE) will be performed in a treadmill while collecting expired gases analysis41. The test will begin at low work rates and gradually increased42 until indications to stop are perceived or volitional exhaustion. The workloads selected for participants should be designed with the aim to reach the maximal effort (peak exercise) in the 8-12 minutes interval43. During CPET maximal oxygen uptake (VO2max) is measured, the stronger predictor of CV risk. It is generally expressed as relative (ml/kg/min)44.
Anthropometric measures | Baseline and 3 months-12 months, every 3 months
  At baseline and at 3, 6, 9, 12 months: weight in kilograms, height in meters, waist circumference, hip circumference, will be measured. Also, BMI Body mass index (BMI): weight in kilograms divided by the square of the height in meters. The cutt-off values are the standards by the WHO97.

CONTACTS AND LOCATIONS:
Overall Officials: Esteban Porrini, MD, PhD, Study Director — Hospital Universitario de Canarias
Locations (1):
- UICEC, San Cristóbal de La Laguna, S/C de TEnerife, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Aktas A. Transplanted kidney function evaluation. Semin Nucl Med. 2014 Mar;44(2):129-45. doi: 10.1053/j.semnuclmed.2013.10.005. PMID 24484750
- [Result] Womer KL, Kaplan B. Recent developments in kidney transplantation--a critical assessment. Am J Transplant. 2009 Jun;9(6):1265-71. doi: 10.1111/j.1600-6143.2009.02639.x. Epub 2009 May 13. PMID 19459815
- [Result] Wolfe RA, Ashby VB, Milford EL, Ojo AO, Ettenger RE, Agodoa LY, Held PJ, Port FK. Comparison of mortality in all patients on dialysis, patients on dialysis awaiting transplantation, and recipients of a first cadaveric transplant. N Engl J Med. 1999 Dec 2;341(23):1725-30. doi: 10.1056/NEJM199912023412303. PMID 10580071
- [Result] Meier-Kriesche HU, Ojo AO, Port FK, Arndorfer JA, Cibrik DM, Kaplan B. Survival improvement among patients with end-stage renal disease: trends over time for transplant recipients and wait-listed patients. J Am Soc Nephrol. 2001 Jun;12(6):1293-1296. doi: 10.1681/ASN.V1261293. PMID 11373354
- [Result] Seoane-Pillado MT, Pita-Fernandez S, Valdes-Canedo F, Seijo-Bestilleiro R, Pertega-Diaz S, Fernandez-Rivera C, Alonso-Hernandez A, Gonzalez-Martin C, Balboa-Barreiro V. Incidence of cardiovascular events and associated risk factors in kidney transplant patients: a competing risks survival analysis. BMC Cardiovasc Disord. 2017 Mar 7;17(1):72. doi: 10.1186/s12872-017-0505-6. PMID 28270107
- [Result] Dahle DO, Grotmol T, Leivestad T, Hartmann A, Midtvedt K, Reisaeter AV, Mjoen G, Pihlstrom HK, Naess H, Holdaas H. Association Between Pretransplant Cancer and Survival in Kidney Transplant Recipients. Transplantation. 2017 Oct;101(10):2599-2605. doi: 10.1097/TP.0000000000001659. PMID 28207636
- [Result] Viecelli AK, Lim WH, Macaskill P, Chapman JR, Craig JC, Clayton P, Cohney S, Carroll R, Wong G. Cancer-Specific and All-Cause Mortality in Kidney Transplant Recipients With and Without Previous Cancer. Transplantation. 2015 Dec;99(12):2586-92. doi: 10.1097/TP.0000000000000760. PMID 26102612
- [Result] Wauters RP, Cosio FG, Suarez Fernandez ML, Kudva Y, Shah P, Torres VE. Cardiovascular consequences of new-onset hyperglycemia after kidney transplantation. Transplantation. 2012 Aug 27;94(4):377-82. doi: 10.1097/TP.0b013e3182584831. PMID 22820698
- [Result] Sharif A, Hecking M, de Vries AP, Porrini E, Hornum M, Rasoul-Rockenschaub S, Berlakovich G, Krebs M, Kautzky-Willer A, Schernthaner G, Marchetti P, Pacini G, Ojo A, Takahara S, Larsen JL, Budde K, Eller K, Pascual J, Jardine A, Bakker SJ, Valderhaug TG, Jenssen TG, Cohney S, Saemann MD. Proceedings from an international consensus meeting on posttransplantation diabetes mellitus: recommendations and future directions. Am J Transplant. 2014 Sep;14(9):1992-2000. doi: 10.1111/ajt.12850. Epub 2014 Aug 6. PMID 25307034
- [Result] Rayburn WF. Diagnosis and classification of diabetes mellitus: highlights from the American Diabetes Association. J Reprod Med. 1997 Sep;42(9):585-6. No abstract available. PMID 9336756
- [Result] Porrini EL, Diaz JM, Moreso F, Delgado Mallen PI, Silva Torres I, Ibernon M, Bayes-Genis B, Benitez-Ruiz R, Lampreabe I, Lauzurrica R, Osorio JM, Osuna A, Dominguez-Rollan R, Ruiz JC, Jimenez-Sosa A, Gonzalez-Rinne A, Marrero-Miranda D, Macia M, Garcia J, Torres A. Clinical evolution of post-transplant diabetes mellitus. Nephrol Dial Transplant. 2016 Mar;31(3):495-505. doi: 10.1093/ndt/gfv368. Epub 2015 Nov 3. PMID 26538615
- [Result] Hagen M, Hjelmesaeth J, Jenssen T, Morkrid L, Hartmann A. A 6-year prospective study on new onset diabetes mellitus, insulin release and insulin sensitivity in renal transplant recipients. Nephrol Dial Transplant. 2003 Oct;18(10):2154-9. doi: 10.1093/ndt/gfg338. PMID 13679495
- [Result] Torres A, Hernandez D, Moreso F, Seron D, Burgos MD, Pallardo LM, Kanter J, Diaz Corte C, Rodriguez M, Diaz JM, Silva I, Valdes F, Fernandez-Rivera C, Osuna A, Gracia Guindo MC, Gomez Alamillo C, Ruiz JC, Marrero Miranda D, Perez-Tamajon L, Rodriguez A, Gonzalez-Rinne A, Alvarez A, Perez-Carreno E, de la Vega Prieto MJ, Henriquez F, Gallego R, Salido E, Porrini E. Randomized Controlled Trial Assessing the Impact of Tacrolimus Versus Cyclosporine on the Incidence of Posttransplant Diabetes Mellitus. Kidney Int Rep. 2018 Jul 11;3(6):1304-1315. doi: 10.1016/j.ekir.2018.07.009. eCollection 2018 Nov. PMID 30450457
- [Result] Hur KY, Kim MS, Kim YS, Kang ES, Nam JH, Kim SH, Nam CM, Ahn CW, Cha BS, Kim SI, Lee HC. Risk factors associated with the onset and progression of posttransplantation diabetes in renal allograft recipients. Diabetes Care. 2007 Mar;30(3):609-15. doi: 10.2337/dc06-1277. PMID 17327329
- [Result] Porrini E, Moreno JM, Osuna A, Benitez R, Lampreabe I, Diaz JM, Silva I, Dominguez R, Gonzalez-Cotorruelo J, Bayes B, Lauzurica R, Ibernon M, Moreso F, Delgado P, Torres A. Prediabetes in patients receiving tacrolimus in the first year after kidney transplantation: a prospective and multicenter study. Transplantation. 2008 Apr 27;85(8):1133-8. doi: 10.1097/TP.0b013e31816b16bd. PMID 18431233
- [Result] Valderhaug TG, Jenssen T, Hartmann A, Midtvedt K, Holdaas H, Reisaeter AV, Hjelmesaeth J. Fasting plasma glucose and glycosylated hemoglobin in the screening for diabetes mellitus after renal transplantation. Transplantation. 2009 Aug 15;88(3):429-34. doi: 10.1097/TP.0b013e3181af1f53. PMID 19667949
- [Result] Luan FL, Langewisch E, Ojo A. Metabolic syndrome and new onset diabetes after transplantation in kidney transplant recipients. Clin Transplant. 2010 Nov-Dec;24(6):778-83. doi: 10.1111/j.1399-0012.2009.01194.x. PMID 20047609
- [Result] Lv C, Chen M, Xu M, Xu G, Zhang Y, He S, Xue M, Gao J, Yu M, Gao X, Zhu T. Influencing factors of new-onset diabetes after a renal transplant and their effects on complications and survival rate. PLoS One. 2014 Jun 9;9(6):e99406. doi: 10.1371/journal.pone.0099406. eCollection 2014. PMID 24911157
- [Result] Al-Ghareeb SM, El-Agroudy AE, Al Arrayed SM, Al Arrayed A, Alhellow HA. Risk factors and outcomes of new-onset diabetes after transplant: single-centre experience. Exp Clin Transplant. 2012 Oct;10(5):458-65. doi: 10.6002/ect.2012.0063. Epub 2012 Aug 29. PMID 22943190
- [Result] Woodward RS, Schnitzler MA, Baty J, Lowell JA, Lopez-Rocafort L, Haider S, Woodworth TG, Brennan DC. Incidence and cost of new onset diabetes mellitus among U.S. wait-listed and transplanted renal allograft recipients. Am J Transplant. 2003 May;3(5):590-8. doi: 10.1034/j.1600-6143.2003.00082.x. PMID 12752315
- [Result] Sharif A, Baboolal K. Risk factors for new-onset diabetes after kidney transplantation. Nat Rev Nephrol. 2010 Jul;6(7):415-23. doi: 10.1038/nrneph.2010.66. Epub 2010 May 25. PMID 20498675
- [Result] Montori VM, Basu A, Erwin PJ, Velosa JA, Gabriel SE, Kudva YC. Posttransplantation diabetes: a systematic review of the literature. Diabetes Care. 2002 Mar;25(3):583-92. doi: 10.2337/diacare.25.3.583. PMID 11874952
- [Result] Knowler WC, Barrett-Connor E, Fowler SE, Hamman RF, Lachin JM, Walker EA, Nathan DM; Diabetes Prevention Program Research Group. Reduction in the incidence of type 2 diabetes with lifestyle intervention or metformin. N Engl J Med. 2002 Feb 7;346(6):393-403. doi: 10.1056/NEJMoa012512. PMID 11832527
- [Result] Pan XR, Li GW, Hu YH, Wang JX, Yang WY, An ZX, Hu ZX, Lin J, Xiao JZ, Cao HB, Liu PA, Jiang XG, Jiang YY, Wang JP, Zheng H, Zhang H, Bennett PH, Howard BV. Effects of diet and exercise in preventing NIDDM in people with impaired glucose tolerance. The Da Qing IGT and Diabetes Study. Diabetes Care. 1997 Apr;20(4):537-44. doi: 10.2337/diacare.20.4.537. PMID 9096977
- [Result] Karamanakos G, Costa-Pinel B, Gilis-Januszewska A, Velickiene D, Barrio-Torrell F, Cos-Claramunt X, Mestre-Miravet S, Piwonska-Solska B, Hubalewska-Dydejczyk A, Tuomilehto J, Liatis S, Makrilakis K. The effectiveness of a community-based, type 2 diabetes prevention programme on health-related quality of life. The DE-PLAN study. PLoS One. 2019 Oct 11;14(10):e0221467. doi: 10.1371/journal.pone.0221467. eCollection 2019. PMID 31603914
- [Result] Didsbury M, McGee RG, Tong A, Craig JC, Chapman JR, Chadban S, Wong G. Exercise training in solid organ transplant recipients: a systematic review and meta-analysis. Transplantation. 2013 Mar 15;95(5):679-87. doi: 10.1097/TP.0b013e31827a3d3e. PMID 23364480
- [Result] Karelis AD, Hebert MJ, Rabasa-Lhoret R, Rakel A. Impact of Resistance Training on Factors Involved in the Development of New-Onset Diabetes After Transplantation in Renal Transplant Recipients: An Open Randomized Pilot Study. Can J Diabetes. 2016 Oct;40(5):382-388. doi: 10.1016/j.jcjd.2015.08.014. Epub 2015 Dec 2. PMID 26656280
- [Result] Sharif A, Moore R, Baboolal K. Influence of lifestyle modification in renal transplant recipients with postprandial hyperglycemia. Transplantation. 2008 Feb 15;85(3):353-8. doi: 10.1097/TP.0b013e3181605ebf. PMID 18301331
- [Result] Abstracts of the 50th ERA-EDTA (European Renal Association-European Dialysis and Transplant Association) Congress. May 18-21, 2013. Istanbul, Turkey. Nephrol Dial Transplant. 2013 May;28 Suppl 1:i1-553. No abstract available. PMID 23682400
- [Result] Dominguez-Rodriguez A, Abreu-Gonzalez P, Mendez-Vargas C, Martin-Cabeza M, Gonzalez J, Garcia-Baute Mdel C, de la Rosa A, Laynez-Cerdena I. Ventilatory efficiency predicts adverse cardiovascular events in asymptomatic patients with severe aortic stenosis and preserved ejection fraction. Int J Cardiol. 2014 Dec 20;177(3):1116-8. doi: 10.1016/j.ijcard.2014.08.073. Epub 2014 Aug 16. No abstract available. PMID 25168095
- [Result] Guazzi M, Arena R, Halle M, Piepoli MF, Myers J, Lavie CJ. 2016 Focused Update: Clinical Recommendations for Cardiopulmonary Exercise Testing Data Assessment in Specific Patient Populations. Circulation. 2016 Jun 14;133(24):e694-711. doi: 10.1161/CIR.0000000000000406. Epub 2016 May 2. PMID 27143685
- [Result] Balady GJ, Arena R, Sietsema K, Myers J, Coke L, Fletcher GF, Forman D, Franklin B, Guazzi M, Gulati M, Keteyian SJ, Lavie CJ, Macko R, Mancini D, Milani RV; American Heart Association Exercise, Cardiac Rehabilitation, and Prevention Committee of the Council on Clinical Cardiology; Council on Epidemiology and Prevention; Council on Peripheral Vascular Disease; Interdisciplinary Council on Quality of Care and Outcomes Research. Clinician's Guide to cardiopulmonary exercise testing in adults: a scientific statement from the American Heart Association. Circulation. 2010 Jul 13;122(2):191-225. doi: 10.1161/CIR.0b013e3181e52e69. Epub 2010 Jun 28. No abstract available. PMID 20585013
- [Result] Obesity: preventing and managing the global epidemic. Report of a WHO consultation. World Health Organ Tech Rep Ser. 2000;894:i-xii, 1-253. PMID 11234459
- [Result] Fauziana R, Jeyagurunathan A, Abdin E, Vaingankar J, Sagayadevan V, Shafie S, Sambasivam R, Chong SA, Subramaniam M. Body mass index, waist-hip ratio and risk of chronic medical condition in the elderly population: results from the Well-being of the Singapore Elderly (WiSE) Study. BMC Geriatr. 2016 Jun 18;16:125. doi: 10.1186/s12877-016-0297-z. PMID 27315800
- [Result] Nishida C, Ko GT, Kumanyika S. Body fat distribution and noncommunicable diseases in populations: overview of the 2008 WHO Expert Consultation on Waist Circumference and Waist-Hip Ratio. Eur J Clin Nutr. 2010 Jan;64(1):2-5. doi: 10.1038/ejcn.2009.139. Epub 2009 Nov 25. PMID 19935820
- [Result] Bushman B. Promoting exercise as medicine for prediabetes and prehypertension. Curr Sports Med Rep. 2014 Jul-Aug;13(4):233-9. doi: 10.1249/JSR.0000000000000066. PMID 25014388
- [Result] Wahid A, Manek N, Nichols M, Kelly P, Foster C, Webster P, Kaur A, Friedemann Smith C, Wilkins E, Rayner M, Roberts N, Scarborough P. Quantifying the Association Between Physical Activity and Cardiovascular Disease and Diabetes: A Systematic Review and Meta-Analysis. J Am Heart Assoc. 2016 Sep 14;5(9):e002495. doi: 10.1161/JAHA.115.002495. PMID 27628572
- [Result] Colberg SR, Sigal RJ, Yardley JE, Riddell MC, Dunstan DW, Dempsey PC, Horton ES, Castorino K, Tate DF. Physical Activity/Exercise and Diabetes: A Position Statement of the American Diabetes Association. Diabetes Care. 2016 Nov;39(11):2065-2079. doi: 10.2337/dc16-1728. No abstract available. PMID 27926890
- [Result] Garber CE, Blissmer B, Deschenes MR, Franklin BA, Lamonte MJ, Lee IM, Nieman DC, Swain DP; American College of Sports Medicine. American College of Sports Medicine position stand. Quantity and quality of exercise for developing and maintaining cardiorespiratory, musculoskeletal, and neuromotor fitness in apparently healthy adults: guidance for prescribing exercise. Med Sci Sports Exerc. 2011 Jul;43(7):1334-59. doi: 10.1249/MSS.0b013e318213fefb. PMID 21694556
- [Result] Thompson PD, Arena R, Riebe D, Pescatello LS; American College of Sports Medicine. ACSM's new preparticipation health screening recommendations from ACSM's guidelines for exercise testing and prescription, ninth edition. Curr Sports Med Rep. 2013 Jul-Aug;12(4):215-7. doi: 10.1249/JSR.0b013e31829a68cf. No abstract available. PMID 23851406
- [Result] Gordon BA, Benson AC, Bird SR, Fraser SF. Resistance training improves metabolic health in type 2 diabetes: a systematic review. Diabetes Res Clin Pract. 2009 Feb;83(2):157-75. doi: 10.1016/j.diabres.2008.11.024. Epub 2009 Jan 9. PMID 19135754
- [Result] Ramachandran A, Snehalatha C, Mary S, Mukesh B, Bhaskar AD, Vijay V; Indian Diabetes Prevention Programme (IDPP). The Indian Diabetes Prevention Programme shows that lifestyle modification and metformin prevent type 2 diabetes in Asian Indian subjects with impaired glucose tolerance (IDPP-1). Diabetologia. 2006 Feb;49(2):289-97. doi: 10.1007/s00125-005-0097-z. Epub 2006 Jan 4. PMID 16391903
- [Result] Kosaka K, Noda M, Kuzuya T. Prevention of type 2 diabetes by lifestyle intervention: a Japanese trial in IGT males. Diabetes Res Clin Pract. 2005 Feb;67(2):152-62. doi: 10.1016/j.diabres.2004.06.010. PMID 15649575
- [Derived] Morales Febles R, Marrero Miranda D, Jimenez Sosa A, Gonzalez Rinne A, Cruz Perera C, Rodriguez-Rodriguez AE, Alvarez Gonzalez A, Diaz Martin L, Negrin Mena N, Acosta Sorensen C, Perez Tamajon L, Rodriguez Hernandez A, Gonzalez Rinne F, Dorta Gonzalez A, Ledesma Perez E, Gonzalez Delgado A, Dominguez-Rodriguez A, Garcia Baute MDC, Torres Ramirez A, Porrini E. Exercise and Prediabetes After Renal Transplantation (EXPRED-I): A Prospective Study. Sports Med Open. 2023 May 18;9(1):32. doi: 10.1186/s40798-023-00574-8. PMID 37202497